CLINICAL TRIAL: NCT06584994
Title: Investigating Clonal Dynamics in Gonads and Their Role in Disease Predisposition
Brief Title: Investigating the Role of Genetics in Disease Predisposition
Status: Enrolling by invitation | Type: Observational
Sponsor: The Wellcome Sanger Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 273194
Record Dates: First submitted 2024-07-04; First posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-07

CONDITIONS: Predisposition, Genetic; Cancer; Mutation; Fertility Disorders
MeSH Terms: conditions — Genetic Predisposition to Disease; Neoplasms | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Extracted DNA, tumour, blood, saliva, buccal samples, skin, semen and human tissue will be stored at Sanger for the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Individuals and Families affected by disease predisposition syndromes: We will work with collaborators to identify cohorts of families in which one or more members suffer with a cancer predisposition syndromes such as LFS. The affected individual/s act as an index participant and their unaffected family members act as controls. This may include immediate family (father, mother and affected/non-affected siblings) and extended family members (grandparents, maternal/paternal uncles and aunts) where practical.
  We wish to collect blood samples, buccal swabs, skin swabs, saliva and/ or urine samples. Adult males (affected and unaffected) may (cohort dependant) also be asked to collect a semen sample for use in the study.
  We will ask affected individuals if we can access any leftover tumour biopsies and/or material from medical procedures for use in the study.Material will only be accessed once it is not required for diagnostic purposes.
  Interventions: Other: sample collection
- Individuals attending fertility clinics with or without fertility problems: For males who are attending fertility clinics we will require blood or saliva samples along with a semen sample as a minimum to take part in this arm of the study.
  Interventions: Other: sample collection
- Individuals receiving treatment for cancers in the reproductive system: These participants will have to agree to donate a blood sample (and a semen sample for adult male participants) both before and after their treatment. If any participants do not wish to give a blood sample, we may be able to collect a saliva sample or buccal swab instead.
  Interventions: Other: sample collection

INTERVENTIONS:
Other: sample collection — Collection of blood, skin, semen, urine and/or saliva samples. Access to previously collected tissue samples (if applicable).

SUMMARY:
Gametogenesis is the production of sperm and eggs; it takes place through the process of meiosis. Gametogenesis is subject to the acquisition of mutations as with other processes in the body. Many of these mutations are somatic, meaning that they occur during life as part of the process of cell division rather than being passed down from parents. When somatic mutations take place during gametogenesis, there is the potential for hereditary genetic consequences. However, the processes that cause the mutations during gametogenesis and the implications they have for heritability and disease predisposition are poorly understood.

The goal of this research is to provide a detailed description of the genetic changes in gonadal tissues, and to understand how mutations acquired during the production of germ cells (sperm and eggs) contribute to the predisposition to a wide range of rare diseases and cancer predisposition in future offspring.

DETAILED DESCRIPTION:
Predisposition to rare disorders and cancers can arise due to mutations (changes in DNA) of sperm cells from father and/or eggs from mother. De novo mutations are genetic alterations that are present for the first time in one family member as a result of a variant (or mutation) in a germ cell (egg or sperm) of one of the parents, or a variant that arises in the fertilized egg itself during early embryogenesis.

Current knowledge about how changes in the sperm and eggs of parents can be inherited by children, is based on genetic sequence analysis of blood from nuclear families. This involved comparison of the changes in DNA of children with that of their parents. Changes that are not present in the blood of parents are likely to have occurred in the sperm and egg of the father and mother.

Whilst studying the nuclear family is very useful in order to look at the level of diversity, it will only allow the investigators to study a small number of germ cells making it difficult to ascertain the overall level of diversity that is shown in the sperm and eggs of fathers and mothers. There is also little knowledge of how different factors such as ageing, smoking, BMI and exposure to carcinogens might affect the germ cells of adults and since changes in sperm and eggs can be transmitted to children, it is important to understand how disease causing mutations arise in reproductive tissues. Thus, how such changes can predispose children to rare disorders and cancer predisposition syndromes.

Previous studies have shown that the FGFR3 gene accumulates more mutations in normal testes during the natural ageing process which leads to the relative enrichment of mutated sperm over time. In rare cases, it can lead to testicular cancer (spermatocytic seminomas) in older men, but also it increases the likelihood of having children with Achondroplasia, which is caused by mutations in the FGFR3 gene in the sperm of the father.

Hence, the investigators aim is to determine the effect of different factors on the recurrence risk of pathogenic (disease causing) mutations in eggs and sperm.

ELIGIBILITY:
Inclusion criteria:

* Minimum of child affected with cancer pre-disposition syndromes and their father
* Additional family members of consented father and child duos (Mother, same parent siblings, Maternal/Paternal Aunts, uncles and grandparents of affected child)
* Reproductive tissue samples from both men and women affected by cancer collected with consent for use in research.
* Reproductive tissue samples from both men and women unaffected by cancer collected with consent for use in research.

Exclusion:

* Fathers who do not wish to donate a semen sample or are unable to will be excluded from the study, as will their families
* Fathers who have had a vasectomy will be excluded from the study as will their families
* Adults who do not have the capacity to consent for themselves will be excluded from the study.
* Families in which both parents do not have capacity to consent will also be excluded as they will be unable to give parental consent for their children's participation.
* In order to be eligible siblings must share the same two parents as the affected child, all other siblings will be excluded from the study.
* Male relatives in the extended family (Maternal/Paternal Aunts, uncles and grandparents of affected child) unwilling or unable to donate both a blood or saliva sample and a semen sample will be excluded from the study.
* Participants who do not have a good understanding of the English language will be excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children diagnosed with disease predisposition syndromes and/or cancer and their family members (mother, father, siblings)
  We may also include the wider family (maternal/paternal aunts, uncles and grandparents)
  Recruitment and the sequencing of both prospectively collected samples and those retrospectively collected from tissue banks will run for the first four years of the study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-06-20 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
How often mutations accumulate in healthy reproductive tissues | 7 years
  Establish how often mutations (changes in DNA) accumulate in healthy reproductive tissues (testes and ovaries).

SECONDARY OUTCOMES:
Identification and Characterisation of Mutations | 7 years
  Determine the genetic changes in gonadal tissues, including the frequency, type, and nature of mutations acquired during germ cell production, and identify the genes and cellular processes that these mutations may alter.
Comparative Analysis of Mutation Rates | 7 years
  Compare mutation rates in gonadal tissues across different age groups, sexes, and individuals with or without cancer predisposition syndromes.
Inheritance and Transmission Risk | 7 years
  Assess the inheritance risk and rate of transmission of pathogenic mutations by analysing the proportion of germ cells carrying these mutations in affected individuals and comparing them to unaffected donors.

CONTACTS AND LOCATIONS:
Overall Officials: Raheleh Rahbari, Principal Investigator — Wellcome Sanger Institute
Locations (1):
- Wellcome Sanger Institute, Cambridge, United Kingdom